CLINICAL TRIAL: NCT01883505
Title: A Phase 2a Multicentre Randomized Double Blind Placebo Controlled Study Followed by an Open Label Period, to Evaluate the Safety, Tolerability and Levodopa Pharmacokinetics in Levodopa-treated Parkinson's Disease Patients With Motor Fluctuations, Administered With Repeated Continuous Subcutaneous ND0612
Brief Title: A Phase 2a Study Followed to Evaluate the Safety, Tolerability and Levodopa Pharmacokinetics in Levodopa-treated Parkinson's Disease Patients Receiving ND0612
Acronym: ND0612/003
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NeuroDerm Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ND0612/003
Record Dates: First submitted 2013-06-09; First posted 2013-06-21 (Estimated); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Parkinson's Disease
Keywords: Motor fluctuations; levodopa pharmacokinetics; levodopa and carbidopa solution; continuous subcutaneous delivery; Patch-pump
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination; Levodopa; Carbidopa; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ND0612 (Experimental): levodopa and carbidopa solution
  Interventions: Drug: Levodopa and carbidopa
- Placebo (Placebo Comparator): Saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levodopa and carbidopa — Subcutaneous continuous administration
  Other Names: Levodopa and carbidopa or saline
  Arms: ND0612
Drug: Placebo — Subcutaneous continuous administration
  Other Names: Saline
  Arms: Placebo

SUMMARY:
This phase 2a randomized double blind placebo controlled, in 30 Parkinson's disease (PD) subjects who are treated with oral levodopa/carbidopa (LD/CD) and suffer from motor fluctuations. The aim of the study is to determine the safety, tolerability, the levodopa pharmacokinetics, the need for oral LD dose adjustment and the usability of the ambulatory drug delivery pump following repeated dosing of ND0612 in a conventional home setting in Parkinson's disease patients. Safety and tolerability, pharmacokinetic profile of levodopa and carbidopa, pump usability and the potential clinical effect of ND0612 will be explored in subjects with PD and motor fluctuations.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women with idiopathic Parkinson's disease
2. Subjects must experience motor fluctuations associated with LD/CD dosing
3. Modified Hoehn and Yahr stage < 5
4. Subjects must be taking optimized and stable levodopa/dopa decarboxylase inhibitor therapy
5. Subjects who are treated with dopaminergic agonists and other anti-PD drugs should be on stable doses
6. Women must be postmenopausal, surgically sterilized, or using adequate birth control. Women of childbearing potential must have a negative pregnancy test (serum beta-HCG) at screening.
7. Subjects must be age 30 or older.
8. Subjects must be willing and able to give informed consent

Exclusion Criteria:

1. Subjects treated with entacapone, tolcapone, stalevo or controlled release formulation of levodopa/carbidopa.
2. Subjects with a clinically significant or unstable medical or surgical condition
3. History of melanoma or significant skin disorders
4. Subjects with significant cognitive impairment
5. Subjects treated with unstable doses of dopaminergic agonists, anticholinergics, Monoamine oxidase (MAO)-B inhibitors, or antipsychotics
6. Subjects with clinically significant psychiatric illness
7. Subjects with a history of alcohol or substance abuse
8. Subjects who have taken experimental medications within 60 days prior to baseline.
9. Subject who have undergone a neurosurgical intervention for Parkinson's disease (e.g., pallidotomy, thalamotomy, transplantation and deep brain stimulation).
10. Subjects with severe disabling dyskinesias.
11. Subjects with hearing, visual or motor impairments that prevent them from using the pump or reacting effectively to errors

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01-06 (Actual); Primary Completion 2015-04-26 (Actual); Study Completion 2015-04-26 (Actual)

PRIMARY OUTCOMES:
Safety | 14 days
  1. Incidence and frequency of adverse events, of dopaminergic adverse events 2. Adverse events reporting related to the ND0612 subcutaneous administration, Draize score 3. Vital signs, physical exam, Laboratory measurements
Levodopa pharmacokinetics (LD PK) | 1hr and 2hr predose, 0h, 0.5 hr, 1hr, 1.5hr, 2hr, 3hr, 4hr, 5hr, 6hr, 7hr, 8hr, 9hr and 10hr hours post oral LD dose
  LD PK parameters: Cmax, Area under the Curve (AUC), T>1000ng/ml, through levels at baseline and during treatment at 14 days.
Tolerability | 14 days
  Withdrawal rates and discontinuations due to adverse events

SECONDARY OUTCOMES:
LD dose adjustment | 14 days
  Change in oral LD total daily dose, change in number of oral LD doses during the first 2 weeks, use of rescue therapy during the third week.
Pump Usability | 14 days
  Simulated usability study, formative Pump usability evaluation. Human factor study. Training on the use of the pump will be performed and questionnaire will be filled to assess the ease of use of the pump and the efficiency of the training.

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Tel Aviv Medical Center, Tel Aviv